CLINICAL TRIAL: NCT01103271
Title: Harnessing the Placebo Effect in Major Depressive Disorder
Brief Title: Pilot Study of Open-label Placebo to Treat Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Director, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2009p002469; K24AT004095 (NIH)
Record Dates: First submitted 2010-04-09; First posted 2010-04-14 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; placebo effect; complementary therapies; alternative therapies
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open-label Placebo Immediate Treatment (Experimental): Participants will begin taking placebo pills for four weeks immediately after enrolling in the study.
  Interventions: Other: Open-label Placebo
- Open-label Placebo Waitlist Treatment (Placebo Comparator): Participants will wait two weeks after enrolling in the study to begin taking placebo pills for four weeks.
  Interventions: Other: Open-label Placebo

INTERVENTIONS:
Other: Open-label Placebo — Participants take open-label placebo pills - two twice daily for four weeks.

SUMMARY:
Placebo pills (pills with no active ingredients) have been shown in research studies to somehow produce self-healing processes. The purpose of this study is to determine whether people will be willing to enter an open-label non-deceptive placebo treatment for Major Depressive Disorder (MDD) and whether open-label placebo can be effective for treating MDD in the context of a supportive physician-patient relationship.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-60 years old.
* Current Major Depressive Disorder (MDD)

Exclusion Criteria:

* Pregnant women or women of child bearing potential not using a medically accepted means of contraception.
* Patients who are a serious suicide or homicide risk.
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* The following Diagnostic and Statistical Manual of Mental Disorders-IV diagnoses: 1) organic mental disorders; 2) substance use disorders, including alcohol, active within the last year; 3) schizophrenia; 4) delusional disorder; 5) psychotic disorders not elsewhere classified; 6) bipolar disorder; 7) acute bereavement; 9) severe borderline or antisocial personality disorder; 10) current primary diagnoses of panic disorder, social phobia, generalized anxiety disorder (GAD), or obsessive compulsive disorder (OCD) (disorders that present as chief complaint and/or have their onset preceding the onset of major depressive disorder).
* Uncontrolled seizure disorder.
* Patients with mood congruent or mood incongruent psychotic features.
* Current use of other psychotropic drugs. Exception: Patients who have been on a stable dose for 30 days of classes of medications such as non-benzodiazepine sedatives, anxiolytic benzodiazepines, non-narcotic analgesics may be included. Flexibility will be allowed based on physician discretion.
* Clinical or laboratory evidence of hypothyroidism.
* Patients who have taken an investigational psychotropic drug within the last year.
* Patients who have not responded to two or more antidepressant trials of adequate doses (e.g., fluoxetine 40 mg/day or higher) and duration (e.g.,for six weeks or more) over the past five years.
* Any concomitant form of psychotherapy (depression focused)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 participants were screened for this study.
Groups:
- Immediate Treatment: Participants will begin taking placebo pills for four weeks immediately after enrolling in the study.
- Waitlist Treatment: Participants will wait two weeks after enrolling in the study to begin taking placebo pills for four weeks.
Period: Overall Study
Arm/Group | Immediate Treatment | Waitlist Treatment
Started | 11 | 9
Completed | 10 | 5
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Waitlist Treatment | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.2 (12.0) | 40.8 (13.7) | 38.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: The primary outcome measure is feasibility, which was operationalized as the number of in-person screens for this study.
Time Frame: One year
Population: The number of participants analyzed is the number of participants screened.
Measure: Number; unit: screens
Groups:
- Placebo Effect Study: These were all participants who were screened for the study but not yet enrolled.
Arm/Group | Placebo Effect Study
Number analyzed (Participants) | 33
screens | 33 (0)

2. Secondary Outcome: Pre-Post Efficacy
Description: The magnitude of the pre-post effect across 4 weeks of treatment, as measured by the Hamilton Rating Scale for Depression-17 (HAMD-17). The HAMD-17 measures depression severity, and has a minimum value of 0 and a maximum value of 52 units on a scale, where higher scores indicate more severe depression.
Time Frame: Screen and 4 weeks (immediate treatment); Baseline and 4 weeks (waitlist treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label-Placebo: Immediate Treatment: Participants assigned to immediate treatment will begin taking placebo pills for four weeks immediately after enrolling in the study.
- Placebo Comparator: Waitlist Treatment: Participants will wait two weeks after enrolling in the study to begin taking placebo pills for four weeks.
Arm/Group | Open Label-Placebo: Immediate Treatment | Placebo Comparator: Waitlist Treatment
Number analyzed (Participants) | 11 | 9
units on a scale | 14.75 (6.61) | 3.25 (6.01)

ADVERSE EVENTS:
Arm/Group | Immediate Treatment | Waitlist Treatment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No